CLINICAL TRIAL: NCT06836921
Title: WECARE APD: Randomized Trial to Evaluate the Impact of a Single Multidisciplinary Team Visit for Atypical Parkinsonian Disorders: a Feasibility Study
Brief Title: WECARE APD: Assessing a Single Multidisciplinary Team Visit for Atypical Parkinsonian Disorders
Acronym: WECARE APD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Deepa Dash, Assistant Professor, Western University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 124694
Record Dates: First submitted 2025-01-29; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Plus
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidisciplinary clinic visit arm (Experimental): The multidisciplinary clinic visit will follow a shared appointment model and involve a specialized team consisting of a movement disorder neurologist, a palliative and critical care neurologist, a cognitive neurologist, a specialist nurse, a physiotherapist, an occupational therapist, a speech-language pathologist, and a social worker. Care will be provided in an outpatient setting at a University Hospital. Before the initial visit, patients with APS and their care partners will complete a pre-visit questionnaire to identify their top three care priorities. During the visit, the multidisciplinary team will meet with the patient and their care partner in a single appointment room, beginning the session by addressing the identified priority issues. The team will collaboratively discuss management strategies, emphasizing self-management, and provide real-time guidance and recommendations. If needed, hands-on physiotherapy and occupational therapy evaluations will be conducted during the
- Waitlist arm (Other): Participants in the control group will receive usual care, consisting of regular management by their neurologist, family physician, and other healthcare providers. This standard care may include referrals to community services, allied health professionals, and other support typically provided during the waitlist period for MDC visit.
  Interventions: Other: Standard of Care (Investigator Choice)

INTERVENTIONS:
Other: Standard of Care (Investigator Choice) — Participants in the control group will receive usual care, consisting of regular management by their neurologist, family physician, and other healthcare providers. This standard care may include referrals to community services, allied health professionals, and other support typically provided during the waitlist period for MDC visit.
  Arms: Waitlist arm
Other: MDC visit — The multidisciplinary clinic visit will use a shared appointment model and will include a specialized team comprising movement disorder neurologist, a palliative and critical care neurologist, a cognitive neurologist, a specialist nurse, a physiotherapist (PT), an occupational therapist (OT), a speech-language pathologist, and a social worker. Care will be delivered in an outpatient setting at a University Hospital. Prior to the initial visit, patients with APS and their care partners will receive a pre-visit questionnaire to identify their top three care priorities.
  During the visit, the multidisciplinary team will convene with the patient and their care partner in a single appointment room. The session will begin by addressing each of the priority issues identified by the patient and care partner. The team will collaboratively discuss management strategies, focusing on self-management, and will provide real-time guidance and recommendations. As indicated, hands-on PT and OT evaluatio

SUMMARY:
Atypical Parkinsonian disorders (APD) are a group of brain disorders that look like Parkinson's disease but progress faster and don't respond well to common treatments like levodopa. These conditions include Progressive Supranuclear Palsy (PSP), Corticobasal Syndrome (CBS), and Multiple System Atrophy (MSA). Caring for APD patients is especially challenging because the symptoms worsen quickly and require multiple specialists, often leading to separate visits with different doctors and therapists. This not only increases the burden on patients and caregivers but also results in high medical costs. Despite the serious impact of APD, there is no proven care model that significantly improves the quality of life for patients and their caregivers.

To address this, the investigator team has created a novel type of clinic that brings together a team of specialists in a shared appointment to provide comprehensive care in one visit. This study aims to test whether an early visit with this team, in addition to regular medical care, can improve quality of life, help patients manage their symptoms better, and reduce the stress on caregivers. The investigators will conduct a six-month study with two groups: one will receive the multidisciplinary care visit right away, while the other will continue with regular care and receive the visit after six months. Patients and caregivers will fill out questionnaires about their well-being at the beginning, after one month, and after six months. The study will also measure how practical it is to run this type of clinic, making sure enough people participate, complete the required surveys, and stay in the study.

This will be the first study to test whether a team-based care model is practical and beneficial for APD patients and their caregivers. If successful, it could serve as a foundation for larger studies and potentially improve care for other complex neurological conditions in the future.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following conditions to be eligible for the study):

* Participants must be older than 40 years.
* The participant must meet the standard international consensus criteria for a clinically probable diagnosis of one of the following neurodegenerative conditions:Multiple System Atrophy (MSA);Progressive Supranuclear Palsy (PSP);Cortico-Basal Syndrome (CBS)

Exclusion Criteria (Participants will be excluded if they meet any of the following conditions):

* Severe Physical or Cognitive Limitations:

  * Participants must be able to attend the clinic.
  * Individuals with severe physical disabilities or cognitive impairments that prevent clinic attendance will be excluded.
* Life-Threatening Comorbidities:

  * Participants with severe, advanced medical conditions that significantly impact survival or functional ability will be excluded. These include, but are not limited to:End-stage renal disease (ESRD) requiring dialysis; End-stage congestive heart failure (CHF) with severe functional impairment; Advanced malignancy (such as metastatic cancer or terminal cancer with limited prognosis).
* Living in long-term care, away from the care-partner

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Eligible Participants Willing to be Randomized | From screening to enrollment , 12 months after study start
  Definition: The proportion of eligible participants who consent to randomization in the study.
  Measurement:
  Total number of eligible participants approached for the study. Number of participants who provide informed consent and agree to be randomized.
  Formula:
  Percentage Willing=( Total Eligible Participants Approached Participants Consented and Randomized )×100
Percentage of Participants Completing Outcome Assessment | At 6 months after randomization
  Definition: The proportion of participants who successfully complete all required outcome assessments at designated time points.
  Measurement:
  Tracking the number of participants who complete each outcome assessment. Comparison of completion rates across different study arms.
  Formula:
  Completion Rate=(Participants Who Complete All Required Assessments Total Participants Enrolled)×100
Satisfaction survey (Quantitative) | After 6 months of randomization
  Response Categories (5-point Likert scale):
  Very satisfied Satisfied Neutral Unsatisfied Very unsatisfied
  Analysis Approach:
  Responses will be dichotomized into:
  Satisfied: Very satisfied + Satisfied Not Satisfied: Neutral + Unsatisfied + Very unsatisfied The proportion of participants in each category will be calculated.
  Formula:
  Satisfaction Rate
  =(Satisfied Responses Total Responses)×100

IPD SHARING:
Plan to Share IPD: No